CLINICAL TRIAL: NCT06396468
Title: Emergence Delirium in Pediatric Age Group: Comparison Between Sevoflurane and Intravenous Anesthesia in Hypospadias Repair: A Randomized Clinical Trial
Brief Title: Sevoflurane and Intravenous Anesthesia in Hypospadias Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ramy Mousa, Professor of Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC 28-11-2023
Record Dates: First submitted 2024-04-22; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-02

CONDITIONS: Emergence Delirium; Intravenous Anesthesia; Sevoflurane
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: In group Sevoflurane, anesthesia was maintained with sevoflurane (1-1.2 MAC) with oxygen /air 1:1.
  In group propofol , anesthesia was maintained continuous infusion of 100-400 mcg/kg /min of propofol and fentanyl 0.1 ug / kg/ min with oxygen /air 1:1.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sevoflurane group (Experimental): Anesthesia was maintained with sevoflurane (1-1.2 MAC) with oxygen /air 1:1
  Interventions: Drug: sevoflurane
- Propofol group (Experimental): Anesthesia was maintained continuous infusion of 100-400 mcg/kg /min of propofol and fentanyl 0.1 ug / kg/ min with oxygen /air 1:1
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: sevoflurane — sevoflurane (1-1.2 MAC)
  Other Names: S group
  Arms: sevoflurane group
Drug: propofol — 100-400 mcg/kg /min of propofol
  Other Names: P group
  Arms: Propofol group

SUMMARY:
Emergence agitation (EA), a phenomenon observed at the time of recovery from general anesthesia (GA).The cause of ED appears to be multifactorial in origin. Use of volatile anesthetics, prolonged duration and type of surgery, pain, and rapid emergence are some factors known to increase its incidence

DETAILED DESCRIPTION:
The pathogenesis of postoperative EA is still undefined, but sevoflurane has intrinsic effects that may share in emergence agitation like its different electroencephalogram pattern from halothane, and its degradation to inorganic fluoride ions and compound A which may have a role in the occurrence of EA Sevoflurane now is the inhalational anaesthetic agent of choice for pediatrics, as it is non-pungent, with minimal airway irritation characters, and its cardiac adverse effects are minimal like cardiac depression and dysrhythmias.

Total intravenous anesthesia (TIVA) using propofol and fentanyl appears to have a smooth recovery profile

ELIGIBILITY:
Inclusion Criteria:

* ages 1 to 8 years
* American society of anesthesiologists (ASA) physical status I and II, scheduled for hypospadias repair

Exclusion Criteria:

* children with a history of active airway disease,
* sleep apnoea, developmental delay,
* psychological,
* neurological disorder,
* cardiovascular abnormality or requirement of post-operative ventilation,
* hepatic impairment, and renal insufficiency, with active upper respiratory tract infection

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-26 (Estimated); Study Completion 2024-07-26 (Estimated)

PRIMARY OUTCOMES:
Emergence delirium | 24 hours
  The pediatric anesthesia emergence delirium (PAED) scale. Each must be evaluated as not at all, just a little, quite a bit, very much, or extremely, where the first three items to be scored reversely (4 = not at all, 0 = extremely) while the last two items to be scored regularly.

SECONDARY OUTCOMES:
FLACC | Postoperatively at 24 hours
  The Face, Legs, Activity, Cry, and Consolability scale is a frequently used tool for pain assessment in children, with a total score of 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Saleh, MD, Principal Investigator — Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No